CLINICAL TRIAL: NCT05192642
Title: Comparative Effectiveness Study of Real-world Control of TRK Fusion Positive Cancer With Patients From Larotrectinib (Vitrakvi) Clinical Trials
Brief Title: A Study Called VICTORIA to Learn More About How Well Larotrectinib Works in Adults With TRK Fusion-positive Cancer by Comparing Larotrectinib Data From Clinical Studies With Data of Other Treatments From Actual Practice
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21993
Record Dates: First submitted 2021-12-05; First posted 2022-01-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Solid Tumors Harboring NTRK Fusion
MeSH Terms: interventions — larotrectinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Larotrectinib clinical trial cohort
  Interventions: Drug: Larotrectinib(Vitrakvi, BAY2757556)
- RW external comparator cohort
  Interventions: Drug: Data on other treatments

INTERVENTIONS:
Drug: Larotrectinib(Vitrakvi, BAY2757556) — Clinical trials
  Groups: Larotrectinib clinical trial cohort
Drug: Data on other treatments — Real word data
  Groups: RW external comparator cohort

SUMMARY:
This is an observational study in which patient data from the past of adult people with solid tumors harboring NTRK gene fusion are studied. This study will focus on 5 tumor types which have been at the late stage or have spread to other parts of the body. These 5 tumor types are:

* Non-small-cell-lung cancer
* Colorectal cancer (located in the intestine)
* Thyroid cancer
* Sarcomas (located in the connective tissue like bones or body fat)
* Salivary gland carcinoma

In some people with cancer, the cancer cells have specific changes in their building plans (genes) called NTRK gene fusion. NTRK stands for neurotrophic tyrosine receptor kinase, the specific gene that is changed. Due to this change in the gene, an altered protein known as a TRK fusion protein is made, which can cause cancer cells to grow and survive. While NTRK is the gene, TRK (tropomyosin receptor kinase) is the name of the protein. The specific cancer is therefore also called TRK fusion-positive cancer.

The study drug, larotrectinib works by blocking the altered TRK fusion protein. Larotrectinib is already available in the US, Europe, and in other countries and is approved for doctors to prescribe to patients with TRK fusion cancer.

The main purpose of this study is to learn more about how well larotrectinib works in adults with TRK fusion-positive cancer compared to other treatments. Researchers will compare how long participants who received larotrectninib lived to how long participants who received other treatments lived. To do this, larotrectinib data from past clinical studies will be compared with data on other treatments gathered from different health data sources. The data will cover the time between January 2013 and end of August 2022.

Besides this data collection, no further tests or examinations are planned and no visits are required in this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced stage of disease or metastatic disease.

Exclusion Criteria:

* Patients involved in TRK inhibitor clinical trials will be excluded from RW control cohort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data is collected globally.
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Retrospective analysis from January 2013 to August 2022

SECONDARY OUTCOMES:
Overall Treatment patterns | Retrospective analysis from January 2013 to August 2022

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer, Whippany, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.